CLINICAL TRIAL: NCT03778944
Title: Renal Graft Functional Enhancement During Donor Anesthesia: A Comparative Study of 3 Modalities
Brief Title: Enhancing Renal Graft Function During Donor Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RGFEDDA
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Renal Failure Chronic; Transplant;Failure,Kidney; Anesthesia
Keywords: Mannitol; Dopamine; Perfusion; Renal graft donor; Anesthesia
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Using computer & sealed envelope randomization, patients are assigned to receive either Mannitol [M group; n=20], Dopamine [D group; n=20] or adequate hydration [C group; n=20]
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- M group (Active Comparator): Mannitol infusion
  Interventions: Procedure: Mannitol infusion
- D group (Active Comparator): Dopamine infusion
  Interventions: Procedure: Dopamine infusion
- C group (Active Comparator): Adequate hydration
  Interventions: Procedure: Adequate hydration

INTERVENTIONS:
Procedure: Mannitol infusion — Infusion of Mannitol 20% at a dose of 0.5 mg/kg to the renal graft donor after induction of anesthesia over 15 minutes.
  Arms: M group
Procedure: Dopamine infusion — Infusion of Dopamine at a dose of 4 microg/kg/min to the renal graft donor after induction of anesthesia till ligation of the renal artery.
  Arms: D group
Procedure: Adequate hydration — Infusion of Ringer Acetate at a rate of 15 ml/kg/hr to the renal graft donor after induction of anesthesia till ligation of the renal artery.
  Arms: C group

SUMMARY:
Renal transplantation is now recognized as the treatment of choice for patients with end-stage renal disease. An optimum anesthetic regimen should enhance the function and perfusion of the transplanted kidney. The aim of this study is to assess & compare the effectiveness of 3 different modalities in this respect: Mannitol, Dopamine and adequate hydration.

ELIGIBILITY:
Inclusion Criteria:

* end-stage renal disease, for living-donor kidney transplantation

Exclusion Criteria:

* severe cardiac or hepatic dysfunction
* coagulopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative creatinine clearance | 7 days
  Post-operative creatinine clearance level of the transplanted kidney graft is measured in ml/min

CONTACTS AND LOCATIONS:
Overall Officials: Nazmy E Seif, MD, Study Chair — Kasr Al-Ainy Hospital, Cairo University; Ahmed M Elbadawy, MD, Study Director — Kasr Al-Ainy Hospital, Cairo University
Locations (1):
- Kasr Al-Ainy Hospital, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided